CLINICAL TRIAL: NCT05677711
Title: A Prospective, Observational Study of the Real World Safety and Effectiveness of the Ultimaster Sirolimus Eluting Coronary Stent System in Subjects With Coronary Artery Lesions in All-comer Patients (MASTER Trial)
Brief Title: Safety and Efficacy of the Ultimaster Stent
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Deok-Kyu Cho, Professor, Yonsei University
Other Study IDs: 9-2021-0152
Record Dates: First submitted 2022-12-12; First posted 2023-01-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Drug-eluting Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultimaster: Ultimaster stent
  Interventions: Device: ultimaster

INTERVENTIONS:
Device: ultimaster — Subjects who received Ultimaster stent will be included.

SUMMARY:
Durable polymer was considered to be the cause of a chronic inflammatory response that leadas to impaired endothelialization of the stent strut and subsequently increases the risk of stent thrombosis. Ultimaster stent (Ultimaster, Terumo Corporation, Tokyo, Japan) are thin strut, silorimus-eluting, biodegradable copolymer to completely degrade over 3-4 months.

DETAILED DESCRIPTION:
Drug-eluting stents (DES) significantly improved outcome compared wiht bare-metal stents because of slow-elution of the antiproliferative drug mixed with a polymer coated on the stent surface. However, the polymers used in the first-generation DES were considered to be the cause of a chronic inflammatory response that leadas to impaired endothelialization of the stent strut and subsequently increases the risk of stent thrombosis. One strategy to mitigate this problem is a biodegradable polymer, which dissolves over time and leaves only the metalic struts behind. Ultimaster stent are silorimus-eluting, biodegradable poly DL-lactide-co-caprolactone copolymer (PDLLA+PCL) to completely degrade over 3-4 months and is also made of 80μm thin strut. The aim of the current study is to investigate the efficacy and safety outcomes in patients treated with ultimaster stents in real-world.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 or older
2. Clinical evidence of coronary artery disease, including asymptomatic ischemia, stable angina, and acute coronary syndromes (unstable angina, non-ST-elevation myocardial infarction, ST-elevation myocardial infarction)
3. No restrictions on the number of blood vessels, number of lesions, and length of lesions
4. Those who voluntarily gave written consent to participate in this clinical study

Exclusion Criteria:

1. Life expectancy within 1 year
2. Subjects with known hypersensitivity or contraindications to the following drugs or substances: heparin, aspirin, clopidogrel, prasugrel, ticagrelor
3. If other researchers judge that it is inappropriate to participate in this study

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients treated with Ultimaster® stents
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
target lesion failures (TLF) per 1 year | 12 months
  Number of 1-year TLF are defined as combination of cardiac death, target vascular myocardial infarction, and ischemia-induced target lesion revascularization

SECONDARY OUTCOMES:
Major Cardiac Adverse Events (MACE) in 1 Year | 12 months
  Number of 1-year MACE are defined as combination of summation of death, myocardial infarction, stent thrombosis, composite variable of target lesion revascularization
cardiac deaths per year | 12 months
  Number of cardiac death at 1 year
1-year non-cardiac death | 12 months
  Number of 1-year non-cardiac death
1-year target vessel myocardial infarction | 12 months
  Number of 1-year target vascular myocardial infarction
1-year Number of non-target vascular myocardial infarction | 12 months
  Number of 1-year non-target vascular myocardial infarction
ischemia-induced target lesion revascularization in 1 year | 12 months
  Number of 1-year ischemia-induced target lesion revascularization
non-ischemic target lesion revascularization in 1 year | 12 months
  Number of 1-year non-ischemic target lesion revascularization
acute stent thrombosis within 24 hours, subacute stent thrombosis within 30 days, and late stent thrombosis at 1 year | within 24 hours, within 30 days, and late stent thrombosis at 1 year
  Number of acute certain or probable stent thrombosis within 24 hours, subacute stent thrombosis within 30 days, and late stent thrombosis at 1 year
strokes per year | 12 months
  Number of 1 year ischemic or hemorrhagic stroke
bleeding events per year | 12 months
  Number of 1-year bleeding rate (Bleeding Academic Research Consortium 2-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No